CLINICAL TRIAL: NCT01069627
Title: An Open-label Study to Assess the Anti-tumor Activity of Avastin in Combination With Fotemustine as First-line Therapy in Patients With Metastatic Melanoma
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Fotemustine in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19309
Record Dates: First submitted 2009-12-15; First posted 2010-02-17 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; fotemustine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: fotemustine

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15 mg/kg intravenously on day 1 of every 3 week cycle
Drug: fotemustine — 100 mg/m² intravenously on Days 1, 8, and 15, followed by 4 weeks of rest, then every 21 days up to 4 to 6 cycles

SUMMARY:
This study will investigate the efficacy and safety of bevacizumab + fotemustine in patients with stage IV melanoma, previously untreated with chemo- or immunotherapy for metastatic disease. Patients will receive Avastin (15mg/kg intravenously[IV]) on Day 1 of every 3 week cycle, in combination with fotemustine (100mg/m² IV) on Days 1, 8 and 15, followed by 4 weeks rest, followed by 100mg/m² IV every 3 weeks for 4-6 cycles. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* cutaneous malignant melanoma;
* advanced, inoperable stage IV melanoma;
* measurable and/or evaluable sites of metastases.

Exclusion Criteria:

* prior chemotherapy and/or IFN/IL2 based immunotherapy for metastatic disease;
* prior malignancies within past 5 years, with the exception of cured non-melanoma skin cancer, or in situ cancer of cervix;
* clinically significant cardiovascular disease;
* ongoing treatment with aspirin (>325mg/day) or other medications known to predispose to gastrointestinal ulceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (4):
- Italy (4):
  - Florence
  - Genova
  - Milan
  - Torino

REFERENCES:
- [Derived] Del Vecchio M, Mortarini R, Canova S, Di Guardo L, Pimpinelli N, Sertoli MR, Bedognetti D, Queirolo P, Morosini P, Perrone T, Bajetta E, Anichini A. Bevacizumab plus fotemustine as first-line treatment in metastatic melanoma patients: clinical activity and modulation of angiogenesis and lymphangiogenesis factors. Clin Cancer Res. 2010 Dec 1;16(23):5862-72. doi: 10.1158/1078-0432.CCR-10-2363. Epub 2010 Oct 28. PMID 21030496

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Fotemustine: Cycle 1 (3-week cycle): Participants received bevacizumab 15 milligrams/kilogram (mg/kg) intravenously (IV) on Day 1 and fotemustine 100 mg per square meter (mg/m^2) IV on Days 1, 8, and 15 followed by 1 week off. Cycle 1 was not repeated.
  Cycle 2 (3-week cycle): Participants received bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off. Cycle 2 was not repeated.
  Cycles 3-8 (3-week cycles): Participants received bevacizumab 15 mg/kg IV and fotemustine 100 mg/m^2 IV on Day 1 followed by 2 weeks off. This cycle was repeated every 3 weeks for 4 to 6 cycles.
  Cycles 9 and beyond (3-week cycles): If the previous 6 to 8 cycles were tolerated with no disease progression, then participants received bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off. This cycle was repeated every 3 weeks until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Bevacizumab + Fotemustine
Started | 20
Completed | 0
Not Completed | 20
Not completed — Disease progression | 7
Not completed — Adverse Event | 12
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who signed the informed consent form, were assigned a study patient number, and took at least one dose of each drug of study combination.
Groups:
- Bevacizumab + Fotemustine: Cycle 1 (3-week cycle): Participants received bevacizumab 15 mg/kg IV on Day 1 and fotemustine 100 mg/m^2 IV on Days 1, 8, and 15 followed by 1 week off. Cycle 1 was not repeated.
  Cycle 2 (3-week cycle): Participants received bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off. Cycle 2 was not repeated.
  Cycles 3-8 (3-week cycles): Participants received bevacizumab 15 mg/kg IV and fotemustine 100 mg/m^2 IV on Day 1 followed by 2 weeks off. This cycle was repeated every 3 weeks for 4 to 6 cycles.
  Cycles 9 and beyond (3-week cycles): If the previous 6 to 8 cycles were tolerated with no disease progression, then participants received bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off. This cycle was repeated every 3 weeks until disease progression or unacceptable toxicity.
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR)
Description: The percentage of participants with an objective response, defined as achieving CR or PR, as evaluated by the Response Evaluation Criteria In Solid Tumors (RECIST) criteria. CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target), PR: at least a 30 percent (%) decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: Intent-to-Treat (ITT) Population: all participants who signed the informed consent form and were assigned a study patient number; data for 1 participant were not assessable as the participant was discontinued from the study due to a protocol violation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 20
percentage of participants | 15 [3 to 38]

2. Secondary Outcome: Time to Progression (TTP) - Percentage of Participants With an Event
Description: TTP was defined as the time in days from the date of first study treatment until the date of tumor progression or death. Failure events were defined as occurrence of death or progression of disease. Data for participants who were alive without tumor progression at the end of the study were censured at the end of the observation period.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; data for 1 participant were not assessable as the participant was discontinued from the study due to a protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 19
percentage of participants | 73.68

3. Secondary Outcome: TTP - Time to Event
Description: TTP was defined as the time in days from the of first study treatment until the date of tumor progression or death. Failure events were defined as occurrence of death or progression of disease. Data for participants who were alive without tumor progression at the end of the study were censored at the end of the observation period. Median TTP was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 19
days | 249.00 [122.00 to 726.00]

4. Secondary Outcome: Duration of CR - Percentage of Participants With an Event
Description: Evaluated only for participants whose best overall response was CR. The start date was the date of first documented CR and the end date was defined as the date of first documented progression of disease, or death. Participants who did not experience progression of disease were censored at last tumor assessment date or at maximum follow-up.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a best overall response of CR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 1
percentage of participants | 0

5. Secondary Outcome: Duration of CR - Time to Event
Description: The start date was the date of first documented CR and the end date was defined as the date of first documented progression of disease, or death. Participants who did not experience progression of disease were censored at last tumor assessment date or at maximum follow-up. Median duration of CR was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a CR were included in the analysis
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 1
days | NA [NA to NA] — Complete response was achieved by a single participant who reached confirmed CR during the study period. This participant did not have worsening of his status during the observation period, no failures were observed relative to this endpoint.

6. Secondary Outcome: Duration of Overall Response of CR or PR - Percentage of Participants With an Event
Description: The start date was the date of first documented CR or PR and the end date was defined as the date of first documented progression of disease, or death. Participants who did not experience progression of disease were censored at last tumor assessment date or at maximum follow-up.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a best overall response of CR or PR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 3
percentage of participants | 66.67

7. Primary Outcome: Percentage of Participants With Clinical Benefit of CR, PR, or Stable Disease (SD)
Description: The percentage of participants with an objective response of CR, PR, or SD, as evaluated by RECIST criteria. CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target), PR: at least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD. SD: steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for pregressive disease (PD). The clinical benefit was finally assessed by computing absolute frequencies and percentages participants with best overall tumor response equal to CR, PR, or SD.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 20
percentage of participants | 65 [41 to 85]

8. Secondary Outcome: Duration of Overall Response of CR or PR - Time to Event
Description: The start date was the date of first documented CR or PR and the end date was defined as the date of first documented progression of disease. Participants who did not experience progression of disease were censored at last tumor assessment date or at maximum follow-up. Median duration of CR or PR was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a best overall response of CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 3
days | 324.00 [155.00 to NA] — Number of data points is too small to support the calculation of an upper limit for the 95% confidence interval.

9. Secondary Outcome: Duration of Stable Disease - Percentage of Participants With an Event
Description: Stable disease was defined as achieving CR, PR, or SD. The start date was the date of first documented CR, PR, or SD and the end date was defined as the date of first documented progression of disease, or death. Participants who did not experience progression of disease were censored at last tumor assessment date or at maximum follow-up.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a best overall response of CR, PR, or SD were included in the anlaysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 12
percentage of participants | 58.33

10. Secondary Outcome: Duration of Stable Disease - Time to Event
Description: Stable disease was defined as achieving CR, PR, or SD. The start date was the date of first documented CR, PR, or SD and the end date was defined as the date of first documented progression of disease, or death. Participants who did not experience progression of disease were censored at last tumor assessment date or at maximum follow-up. Median duration of CR, PR, or SD was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a best overall response of CR, PR, or SD were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 12
days | 619.00 [249.00 to NA] — Number of data points is too small to support the calculation of an upper limit for the 95% confidence interval.

11. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the starting day of the therapy up to death or the last date the participant was known to be alive.
Time Frame: Baseline, every 3 weeks to end-of-treatment, every 3 months during follow-up, to death or end-of-study (maximum of 36 months)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 20
percentage of participants | 60

12. Secondary Outcome: OS - Time to Event
Description: The time from the starting day of the therapy up to death or the last date the participant was known to be alive. Median OS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 11
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 20
days | 615.00 [298.00 to 796.00]

13. Secondary Outcome: Time to Treatment Failure (TTF) - Percentage of Participants With an Event
Description: The time from date of start of treatment to the earliest among date of progression, date of death due to any cause, or date of discontinuation due to reason other than 'Protocol Violation' or 'Administrative Problem'. For the participants who did not experience treatment failure, TTF was censored at last adequate tumour assessment.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 19
percentage of participants | 100

14. Secondary Outcome: TTF - Time to Event
Description: The time from date of start of treatment to the earliest among date of progression, date of death due to any cause, or date of discontinuation due to reason other than 'Protocol Violation' or 'Administrative Problem'. For the participants who did not experience treatment failure, TTF was censored at last adequate tumour assessment. Median TTF was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 19
days | 126.00 [43.00 to 158.00]

15. Secondary Outcome: Time to CR - Percentage of Participants With an Event
Description: The time between date of start of treatment until first documented CR. This analysis included all responders. Participants who did not achieve a confirmed CR were censored at last adequate tumour assessment date or at maximum follow-up.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 19
percentage of participants | 5.26

16. Secondary Outcome: Time to CR - Time To Event
Description: The time between date of start of treatment until first documented CR. This analysis included all responders. Participants who did not achieve a confirmed CR were censored at last adequate tumour assessment date or at maximum follow-up. Mean time to CR was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT population; only participants with a CR were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 1
days | 76.00 (NA) — Number of data points is too small to support the calculation of the standard deviation.

17. Secondary Outcome: Time to Overall Response of CR or PR - Percentage of Participants With an Event
Description: The time between date of start of treatment until first documented response of CR or PR. This analysis included all responders. Participants who did not achieve a confirmed CR or PR were censored at last adequate tumour assessment date or at maximum follow-up.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 19
percentage of participants | 15.79

18. Secondary Outcome: Time to Overall Response of CR or PR - Time to Event
Description: The time between date of start of treatment until first documented response of CR or PR. This analysis included all responders. Participants who did not achieve a confirmed CR or PR were censored at last adequate tumor assessment date or at maximum follow-up. Mean time to CR or PR was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks during study treatment, and every 3 months during follow-up, up to 36 months
Population: ITT Population; only participants with a response of CR or PR were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bevacizumab + Fotemustine
Number analyzed (Participants) | 3
days | 116.50 (7.58)

ADVERSE EVENTS:
Time Frame: From date of first administration of study drug to 28 days after last administration of study drug.
Arm/Group | Bevacizumab + Fotemustine
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Fotemustine (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Fotemustine (N=20)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Gastric dilatation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oesophageal achalasia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Salivary gland mass (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 10
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 3
Hypersensitivity (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase (Investigations) | 1
Aspartate aminotransferase (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.